CLINICAL TRIAL: NCT02470260
Title: Northern Manhattan Study of Metabolism and Mind
Acronym: NOMEM
Status: Active, not recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, José A. Luchsinger, Professor of Medicine and Epidemiology, Columbia University
Other Study IDs: AAAQ2950; P60MD000206 (NIH); R01AG050440 (NIH)
Record Dates: First submitted 2015-06-08; First posted 2015-06-12 (Estimated); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Diabetes; Pre-diabetes; Cognition - Other; Depressive Symptoms; Metabolic Syndrome
Keywords: Diabetes; Pre-diabetes; Cognition; Depressive symptoms
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Depression; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood for DNA extraction, plasma, sera
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diabetes: Defined by clinical history or HbA1c criteria (HbA1c greater of equal to 6.5%)
- Pre-diabetes: Defined by HbA1c criteria (5.7 to 6.4%)
- Normal glucose tolerance: Defined by HbA1c criteria (< 5.7%)

SUMMARY:
Pre-diabetes, type 2 diabetes, and their related conditions, adiposity and insulin resistance, are more prevalent in minorities Northern Manhattan compared to the general population of the United States. Despite knowledge of the main biologic determinants of these conditions (high caloric intake and sedentarism) the prevalence of these conditions continue to increase. In addition, these conditions can cause mental health problems including increased depressive symptoms and cognitive impairment. Thus, the investigators decided to conduct a community based study of middle aged Hispanic men and women aged 50 to 64 years at baseline in order to:

1. Document the prevalence and incidence, of pre-diabetes, diabetes, overweight, obesity, and associated conditions (e.g. dyslipidemia, hypertension).
2. Study how social determinants of health (SDOH) affect these conditions.
3. Study the consequences of these conditions on aging and mental health outcomes, including cognitive impairment.

DETAILED DESCRIPTION:
DESIGN OVERVIEW: the Northern Manhattan Study of Metabolism and Mind (NOMEM) is a longitudinal cohort study of middle aged Hispanics. Recruitment of the initial cohort of 600 participants was completed between January of 2012 and December of 2013. Our total target sample size is 1000 participants. Participants are followed every 2 years. Participants are self-identified Hispanic men and women aged 50 to 65 years. The sampling frame is the community of Northern Manhattan in New York City.

Participants undergo phlebotomy, measurement of vital signs and anthropometric measures, interviews of medical history, cognitive assessments, and interviews of social determinants of health and mental and physical conditions. Assessments take between 2 and 3 hours.

VARIABLES:

* Glycemia and diabetes status: glycemia is measured with HbA1c. Diabetes is defined by clinical history or by HbA1c ≥ 6.5%, following 2010 ADA criteria. Pre-diabetes is determined following ADA 2010 criteria (HbA1c 5.7 to 6.4%).
* APOE genotyping: The 3 APOE alleles will be genotyped, ε2, ε3, and ε4.
* Body Mass Index (BMI). Standing height is measured using a stadiometer calibrated in cm. Body weight is measured using a balance beam scale calibrated in kg. With the participant standing, measurements are taken to the nearest 0.1 kg of weight with a balance scale and height without shoes to nearest 0.5 cm, to calculate BMI (weight/height2). (use: covariate, ancillary studies).
* Demographic variables: We collect date of birth, sex, years and education, racial group, and country of origin (following the 2010 census format for Hispanics) (use: covariates).
* Depression: We measure depression and depressive symptoms using the PHQ9 and the PROMIS depression scale.
* High sensitivity CRP: Measured using ELISA (Diagnostic systems laboratories, INC, Webster, Texas). The assay sensitivity is 1.6 ng/ml, the inter-assay CV is 11.7%, and the intra-assay CV is 4.6%. This assay can be conducted in serum or plasma.
* Lipids: total cholesterol (TC), HDL. TC and HDL are measured using enzymatic colorimetric methods (Vitros; Johnson & Johnson, New Brunswick, NJ).
* Medical history.This includes vascular disease, cancer, and smoking
* Medications: We will record medications, vitamins, and over the counter products (use: covariate, ancillary studies).
* Resting blood pressure (BP): BP will be measured using an automated oscillometric device; 3 measurements are obtained at 1-minute intervals in a seated position after 5 minutes of rest. The average of the 2nd and 3rd measurements will be recorded as the BP.
* Waist and hip circumference: Waist circumference is measured at the level of the umbilicus. Hip circumference is measured at the level of maximal protrusion of the gluteal muscles. Waist-hip ratio is calculated as the ratio of waist circumference to hip circumference.
* Cognitive battery:

  * WAIS-R Similarities. This Wechsler Adult Intelligence Scale-Revised subtest has good norms and is a standard portion of a dementia evaluation. The items have been translated into Spanish and a scoring guide has been developed. Age-Scaled scores will be used. [Max. Score=19; Time=5 min] Non-Verbal Similarities. The Identities and Oddities subtest of the Mattis Dementia Rating Scale is used to assess nonverbal abstract reasoning. [Max. Score=16; Time=2 min]
  * Color Trails Test Color Trails 1 is a test of sustained visual attention, psychomotor speed, and simple sequencing and involves connecting circles containing the numbers 1 through 25 in order as quickly as possible. Color Trails 2 also involves connecting circles containing the numbers 1 through 25 in order as quickly as possible, but the examinee must shift between pink and yellow colored circles. Like Part 1, Color Trails 2 assesses visual attention and psychomotor speed but also requires a higher level of executive functioning skills.
  * Verbal Fluency: Controlled Word Association Test. The patient is given 1 min to name as many words beginning with a particular letter as s/he can. Norms and frequency counts exist for this test in Spanish as well as English. Three categories, Animals, Food, and Clothing are administered to assess category naming. [Time=7 min]
  * The Selective Reminding Test (SRT) is a standard tool in the assessment of verbal memory and dementia and has been used as a sensitive longitudinal measure of changes in memory function. The SRTwas translated into Spanish using words of similar frequency to those in the standard test versions. Subjects are given 6 trials to learn a list of 12 unrelated words. After each attempt at recalling the list, the subject is reminded only of the words that were not recalled and then must attempt to recall the entire list. To assess short-term memory, 2 measures are used: total recall (max. score=72) and retrieval from long-term storage (max. score=72). To assess long-term recall, delayed recall is assessed 15 minutes after completing the SRT (max. score=12); recognition of words not recalled is then tested using multiple choice arrays (max. score=12). [Time (not including 15 min. delay interval, during which other tests are administered) =15 min].
  * The orientation items from the modified Mini-Mental State Examination are used to assess orientation to time and place. These items are sensitive to dementing changes in our normative samples. [Max. Score=10; Time to administer=2 min]
* Social Determinants of Health:

  * Individual SES: MacArthur Network on SES and Health Measures Household income/number of people supported, wealth, debt, how long one could live at current lifestyle if current sources of income ceased
  * Perceived Social Status: MacArthur Ladder; Perceived relative standing in the US
  * Migration: Age at migration Years of life in US
  * Everyday Discrimination* Everyday Discrimination; 10 items; Daily discriminatory hassles
  * Major Discrimination* Modified Experiences of Discrimination Scale:

    12 items; Frequency measure of total lifetime occurrences; 0=Never to 5=Four or More Times
  * Coping with Discrimination-Psychosocial Experiences of Discrimination Scale; 3 coping styles-0=Passive (accept/quiet); 1=Moderate (quiet); 2=Engaged (do something/talk to others)
  * Coping with Discrimination-Health Behavior Modified Experiences of Discrimination Scale 4 behaviors-Exercising, eating sweets/fatty foods, drinking alcohol, smoking cigarettes 0=Never; 3=most of the time
  * Coping with Stress-Psychosocial Based on Experiences of Discrimination Scale 3 coping styles-0=Passive (accept/quiet); 1=Moderate (quiet); 2=Engaged (do something/talk to others)
  * Coping with Stress-Health Behavior Modified Experiences of Discrimination Scale 4 behaviors-Exercising, eating sweets/fatty foods, drinking alcohol, smoking cigarettes; 0=Never; 3=most of the time
  * Racial/Ethnic Socialization Racial/Ethnic Socialization Scale 15 items; 0=Never, 1=Almost Never; 2=Sometimes; 3=Often; 4=Very Often
  * Ethnic Identity Multi-Ethnic Identity Measure 12 items from Affirmation and Belonging and Ethnic Identity Search subscales
  * Acculturation Bidimensional Acculturation Scale Average of 12 items in each domain (Hispanic, Non-Hispanic)
  * Alcohol Use Alcohol Use Disorders Identification Test 10 items; Items scored 0-4
  * Smoking From COHD battery Cigarettes smoked daily
  * Diet Behavioral Risk Factor Surveillance System 6 items; 1=More than Once a Day; 5=Less than Once a Week
  * Physical Activity IPAQ Summation of the duration (in minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activities to estimate MET minutes/week
  * Barriers to Exercise* Benefits and Barriers to Exercise71 9 items; 0=Never; 5=Very Often
  * John Henryism John Henryism Active Coping Scale 12 items; 1=Completely True; 5=Completely False
  * Social Support Social Support Questionnaire Count # of people for odd items. Add totals (Max=54). Divide by 6 for per item SSQ Number Score. Add total Satisfaction score for 6 even numbered items
  * Neighborhood Resources Census-derived neighborhood deprivation % living or below poverty line

ELIGIBILITY:
Inclusion Criteria:

* Self identified Hispanic (any Hispanic subgroup)
* Man or woman.
* Between the ages of 50 and 64 years at baseline

Exclusion Criteria:

* History of cancer other than non-melanoma skin cancer

  * The expectation of moving out for the country permanently before during the study period
  * Presence of a clinical diagnosis of dementia, which we anticipate will be unlikely in this age group.
  * Visual, hearing, or physical impairment that precludes active participation in the study and inability to complete study questionnaires.

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Middle aged Hispanics from Northern Manhattan, New York City
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cognition | 6 years
  cognitive change over at least 3 follow-ups measured with the Selective Reminding Test, Color trails test, and Animal fluency tests.

SECONDARY OUTCOMES:
Transitions in diabetes status | 6 years
  Transition from a diabetes state (normal glucose tolerance, pre-diabetes, diabetes) to another state (normal glucose tolerance, pre-diabetes,diabetes).
  HbA1 is used to ascertain Normal glucose tolerance (HbA1c < 6.7%) and pre-diabetes (HbA1c between 6.7 and 6.49%).
Metabolic syndrome | 6 years
  The components of the metabolic syndrome are:hyperglycemia (pre diabetes or diabetes), central obesity (determined with waist circumference, low HDL, hypertension, and inflammation (hsCRP > 3); the metabolic syndrome is present when 3 or more of the components are present.
Depressive symptoms | 6 years
  assessed with the PHQ9 and the PROMIS depression scale

CONTACTS AND LOCATIONS:
Overall Officials: Jose A. Luchsinger, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided